CLINICAL TRIAL: NCT06441604
Title: Extended-release Buprenorphine as a Novel Low-dose Induction Strategy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: University of Utah (Other)
Responsible Party: Principal Investigator, Joji Suzuki, MD, Director, Division of Addiction Psychiatry, Brigham and Women's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2024P001078
Record Dates: First submitted 2024-05-08; First posted 2024-06-04 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Opioid Use Disorder
Keywords: Opioid Use Disorder; Buprenorphine
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Intervention Model Description: The study is a single-blind, fixed-order, dose-escalation designed trial in an inpatient setting with individuals with a DSM-5 diagnosis of OUD (n=30). The first 10 participants will receive XR-BUP 16mg in single-blind fashion. We will then proceed with 10 more participants to the 24mg dose, and finally proceed with 10 more participants to the 32mg dose. All participants will receive fentanyl to prevent withdrawal symptoms. (Figure 2). Symptomatic treatments will be provided at any sign of worsening withdrawal including evidence of precipitated withdrawal.
Who Masked: Participant
Masking Description: Only the participant will be masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 16mg Extended-Release Buprenorphine (Experimental): The first 10 participants will receive XR-BUP 16mg in single-blind fashion.
  Interventions: Drug: Extended-release Buprenorphine
- 24mg Buprenorphine (Experimental): After first 10 participants have been completed, the next 10 participants will receive 24mg in a single-blind fashion.
  Interventions: Drug: Extended-release Buprenorphine
- 32mg Buprenorphine (Experimental): After the 20 participants have been completed, the next 10 participants will receive 32mg in a single-blind fashion.
  Interventions: Drug: Extended-release Buprenorphine

INTERVENTIONS:
Drug: Extended-release Buprenorphine — The study is a single-blind, fixed-order, dose-escalation designed trial in an inpatient setting with individuals with a DSM-5 diagnosis of OUD (n=30). The first 10 participants will receive XR-BUP 16mg in single-blind fashion. We will then proceed with 10 more participants to the 24mg dose, and finally proceed with 10 more participants to the 32mg dose. All participants will receive fentanyl to prevent withdrawal symptoms. (Figure 2). Symptomatic treatments will be provided at any sign of worsening withdrawal including evidence of precipitated withdrawal.

SUMMARY:
This is a clinical trial to characterize the safety and pharmacokinetics of using extended-release buprenorphine (XR-BUP) as a novel low-dose buprenorphine induction strategy. Individuals with a diagnosis of Opioid Use Disorder (OUD) (n=30) will be admitted to an inpatient unit to complete study procedures over the course of 3 days. Participants will receive fentanyl to prevent the emergence of withdrawal. Each participant will then receive a single injection of XR-BUP after which study staff will monitor for any precipitated withdrawal.

DETAILED DESCRIPTION:
The approach is to conduct a single ascending dose trial in a controlled human laboratory setting with individuals with a diagnosis of OUD (n=30) actively using illicit fentanyl. After obtaining informed consent and establishing eligibility, 10 participants will be scheduled for an inpatient visit lasting 3 days, 2 nights and receive XR-BUP when not yet experiencing any opioid withdrawal. Participants will receive fentanyl to prevent the emergence of withdrawal, and on the following morning, receive XR-BUP 16mg in single-blind fashion. If at least 90% successfully complete induction (success defined as experiencing no precipitated withdrawal) with the 16mg dose, then we will proceed with 10 more participants to receive the 24mg dose. If at least 90% successfully complete induction the 24mg dose, then we will proceed with 10 more participants to the 32mg dose. Timed blood samples will be collected in heparinized Vacutainer tubes via a catheter in the antecubital vein at baseline, and at 0.5, 1, 2, 4, 6, 8, 12, and 24 hours after the XR-BUP injection.

ELIGIBILITY:
Inclusion Criteria:

* English speaking adults aged 18 and above.
* diagnosis of opioid use disorder.
* Self-reporting use of illicit opioids in >21 days in the prior 30 days.
* Provide urine toxicology testing positive for fentanyl at baseline.

Exclusion Criteria:

* Seeking medication treatment for opioid use disorder with sublingual buprenorphine or methadone.
* Received buprenorphine or methadone treatment in prior 30 days.
* Current diagnosis of alcohol or sedative/hypnotic use disorder.
* Positive urine drug screen for benzodiazepines, alcohol and or methadone.
* Physical dependence on alcohol or sedative/hypnotics.
* Psychotic disorder, active suicidality or homicidally or any psychiatric condition that impair ability to provide informed consent.
* Have a history or diagnosis of Intracranial mass/bleed, seizure disorder, liver cirrhosis, renal failure, obstructive lung disease, hyperthyroidism, narrow-angle glaucoma, valvular heart disease, cardiac arrhythmias, heart failure.
* Recent (within 6 months) head trauma, stroke, or myocardial infarction
* Requiring treatment with opioids for acute or chronic pain.
* History of hypersensitivity or allergy to buprenorphine or fentanyl.
* Pregnant or breastfeeding.
* Liver function test greater than 3 times upper normal limit.
* Receiving medications that are strong or moderate CYP34A inducers or inhibitors (including but not limited to ketoconazole, itraconazole, clarithromycin, fluconazole, erythromycin), in the past 30 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-10-27 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of XR-Buprenorphine | For the duration of the inpatient admission, lasting 24 hours after receipt of study drug.
  The primary outcome is the proportion of participants who successfully complete induction, defined as experiencing no BPOW, which will be assessed using the COWS. An increase in the COWS score by 8 or more with the total score exceeding 13, within 4 hours will be considered BPOW.
Plasma-concentration curves (AUC) of buprenorphine. | Baseline, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours after study drug administration.
  The area under the plasma concentration curves (AUC) of buprenorphine will be determined.
  Timed blood samples will be collected in anticoagulant Vacutainer tubes via venipuncture at baseline, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours after the XR-BUP injection. Samples will be centrifuged and frozen until analysis.

SECONDARY OUTCOMES:
Maximum Plasma Concentration | Baseline, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours after study drug administration.
  Plasma data will be used to calculate maximum plasma concentration (Cmax) for buprenorphine, norbuprenorphine, and their glucuronides.
Minimum Plasma Concentration (Cmin), | Baseline, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours after study drug administration.
  Plasma data will be used to calculate minimum plasma concentration (Cmin) for buprenorphine, norbuprenorphine, and their glucuronides.
Time to Maximum Plasma Concentration | Baseline, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours after study drug administration.
  Plasma data will be used to calculate time to maximum plasma concentration (Tmax) for buprenorphine, norbuprenorphine, and their glucuronides.
Elimination half-life | Baseline, 0.5, 1, 2, 4, 6, 8, 12, and 24 hours after study drug administration.
  Plasma data will be used to calculate elimination half-life (t1/2) for buprenorphine, norbuprenorphine, and their glucuronides.
Buccal Swab | will be done once at the baseline visit.
  DNA testing to check 3A4 activity levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States